CLINICAL TRIAL: NCT03375372
Title: Effects of Periodontal Therapy on Markers of Acute Phase Response (APR), Oxidative Stress: Phase II {Formerly UNC Biomedical IRB Study # DENT-2019}
Brief Title: Effects of Periodontal Therapy on Markers of Acute Phase Response, Oxidative Stress
Acronym: BCU2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-1516
Record Dates: First submitted 2017-12-06; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Treatment Group) (Active Comparator): Subjects receive intervention of Scaling and Root Planing (S&RP) procedure under local anesthesia, plus a specified Oral Hygiene Regimen (OHR)
  Interventions: Procedure: Scaling and Root Planing (S&RP)
- Group 2 (Delayed treatment) (No Intervention): Subjects have delayed treatment scaling and root planing procedure and OHR at 36 weeks (Final visit) These subjects are not followed beyond completion of the treatment.

INTERVENTIONS:
Procedure: Scaling and Root Planing (S&RP) — dental Scaling and Root Planing and oral hygiene regimen
  Other Names: Scaling & Root Planing (S&RP)
  Arms: Group 1 (Treatment Group)

SUMMARY:
This study began enrollment in 2003 with final report completed in October of 2015. This submission is being provided to acquire an NCT number.

This study was successfully executed according to protocol with full enrollment and completion of 89.7% of subjects. Subjects were enrolled into a two arm study 1) Combined therapy (scaling and root planing plus Crest products) vs. 2) delayed treatment. Subjects were followed for 6 months and a wide and extensive battery of biological samples were collected to determine the effects of treatment on the local and systemic inflammatory response.

DETAILED DESCRIPTION:
The design for this study was a single-blinded, delayed treatment, controlled, randomized, clinical trial. A total of 106 subjects, 2 sets of 53 patients each in one of 2 arms, were enrolled. For both groups at 6 weeks, 3 months, and 6 months periodontal measures, gingival crevicular fluid, and plaque were taken using standardized techniques. Blood for serum was collected at each time point, plus at an additional 2 week visit. GCF samples were collected and analyzed for PGE2 and IL-1 to provide a mediator assessment of periodontal status.These GCF data and the clinical changes were used to assure that the therapy provided had resulted in a local therapeutic benefit. These data were primarily useful as it relates to changes in systemic levels of mediators.

Subjects were recruited from the surrounding communities by means of flyer advertisements, as well as media advertisements in weekly newspapers and on the radio. Recruitment focused on subjects between the ages of 18 and 64 years with periodontal disease.

The investigators excluded persons who have less than 20 teeth; who had any serious systemic disease including: auto-immune type disorders (i.e. systemic lupus erythematous), immunosuppression (chronic systemic c steroid use, cancer chemotherapy or HIV infection), chronic liver disease including hepatitis, or diabetes mellitus; extremely obese (BMI <40), are pregnant, or who abuse alcohol or drugs. Subjects were selected from periodontal screening examinations as having 4 or more sites with pocket depths of 5 or more mm and two or more sites with attachment loss of 3 mm or more and who required scaling and root planing.

The Phase II set of 106 patients had periodontal therapy consisting of one of two treatments:

Treatment 1: A 6-week observation period (treatment delay), then full-mouth scaling and root planing plus specific oral hygiene regimen (OHR) (Group 1);

Treatment 2: A 6-week observation period (treatment delay), then a further 6-month observation period (delayed treatment), followed by scaling and root planing plus specific oral hygiene regimen (OHR) at 6 months (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* subjects with four or more periodontal pockets of five millimeters or greater and two or more sites with an clinical attachment loss of three millimeters or greater.

Exclusion Criteria:

* subjects with less than 20 teeth
* subjects with serious systemic diseases (lupus, systemic erythematous), immunosuppression (chronic systemic steroid use, cancer, chemotherapy, or HIV infection), chronic liver disease including hepatitis or diabetes mellitus.
* Body Mass Index of of 40 or greater
* pregnant
* abuse alcohol or drugs

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2003-04-11 (Actual); Primary Completion 2004-08-01 (Actual); Study Completion 2005-06-04 (Actual)

PRIMARY OUTCOMES:
Effects of S&RP & OHR on C-Reactive protein | 6 months post S&RP
  Delta log value pg/ml 6 months post S&RP & OHR
Effects of S&RP & OHR on HDL cholesterol | 6 months post S&RP
  Delta log value mg/dL 6 months post S&RP & OHR
Effects of S&RP & OHR on LDL cholesterol | 6 months post S&RP
  Delta log value mg/dL 6 months post S&RP & OHR
Effects of S&RP & OHR on VLDL cholesterol | 6 months post S&RP
  Delta log value mg/dL post S&RP & OHR
Effects of S&RP & OHR on Triglycerides | 6 months post S&RP
  Delta log value mg/dL 6 months post S&RP & OHR
Effects of S&RP & OHR on sCD-14 | 6 months post S&RP
  Delta log value µg/ml 6 months post S&RP & OHR
Effects of S&RP & OHR on Homocysteine | 6 months post S&RP
  Delta log value μmol/L 6 months post S&RP & OHR
Effects of S&RP & OHR on 8-isoprostane | 6 months post S&RP
  Delta log value pg/ml 6 months post S&RP & OHR
Effects of S&RP & OHR on sICAM | 6 months post S&RP
  Delta log value pg/ml 6 months post S&RP & OHR
Effects of S&RP & OHR on Apolipoprotein A | 6 months post S&RP
  Delta log value mg/dL 6 months post S&RP & OHR

SECONDARY OUTCOMES:
Relationship between S&RP and OHR on PGE2 & IL-1beta | 6 months post S&RP
  to determine the relationship between the effects of S&RP plus OHR on levels of systemic inflammation and local changes in periodontal status, GCF levels of PGE2 and IL-1 and the periodontal microbiota, quantifying the levels of 40 organisms.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS PhD MMsc, Principal Investigator — Chair of UNC Periodontology

IPD SHARING:
Plan to Share IPD: Undecided